CLINICAL TRIAL: NCT00708071
Title: An Exploratory Phase 2 Clinical Study to Evaluate Efficacy and Safety of the Adjuvant Use of Fibrin Sealant With 4 IU/mL Thrombin, Vapor Heated, Solvent Detergent Treated Containing Synthetic Aprotinin (FS VH S/D 4) in Subjects Undergoing Rhytidectomy
Brief Title: Efficacy and Safety Study of Fibrin Sealant With 4 IU/mL Thrombin, Vapor Heated, Solvent Detergent Treated (FS VH S/D 4) in Face-Lift Procedures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 550703
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Facial Rhytidectomy (Face-lift)
MeSH Terms: interventions — Fibrin Tissue Adhesive; Thrombin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): One side of the face is treated with FS VH S/D 4; the other side of the face is treated using standard of care.
  Interventions: Biological: Fibrin Sealant with 4 IU/ml Thrombin, Vapor-Heated, Solvent Detergent Treated Containing Synthetic Aprotinin (FS VH S/D 4)

INTERVENTIONS:
Biological: Fibrin Sealant with 4 IU/ml Thrombin, Vapor-Heated, Solvent Detergent Treated Containing Synthetic Aprotinin (FS VH S/D 4) — Each subject received fibrin sealant with 4 IU/mL thrombin, vapor heated, solvent detergent treated containing synthetic aprotinin (FS VH S/D 4 ) to one side of the face. The dosing volume to be applied is 0.02 mL/cm2 to 0.04 mL/cm2. The study product will be applied to the subcutaneous plane in both the neck and the face area. The product will be applied using the spray device provided by the sponsor. (The other side of the face will be treated using standard of care.)
  Other Names: Fibrin Sealant; TISSEEL

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of fibrin sealant with 4 IU/mL thrombin, vapor heated, solvent detergent treated (FS VH S/D 4) when used to reduce early postoperative bruising in participants undergoing a rhytidectomy (face-lift).

ELIGIBILITY:
Inclusion Criteria:

* Subjects planned for facial rhytidectomy
* Subjects who read, understand and sign the written informed consent
* Healthy female or male subjects as determined by the investigator using standard pre-operative assessments to include laboratory tests and ECG
* Subjects 18-75 years old, inclusively
* Subjects who are able and willing to comply with the protocol requirements
* Female subjects of childbearing potential with a negative urine or serum pregnancy test within 72 hours of surgery

Exclusion Criteria:

* Pregnant or lactating women
* Subjects who have undergone previous face-lift surgery
* Subjects undergoing abbreviated face-lift procedures such as deep plane procedures, minimal undermining procedures, thread lifts, and minimal access cranial suspension
* Subjects indicated for concurrent facial surgeries during the operation (e.g. forehead plasty, blepharoplasty, rhinoplasty, buccal fat removal, any filler injections including fat injections, lip augmentation, skin resurfacing procedures etc.)
* Subjects indicated for additional procedures during the same operation (e.g., liposuction, mastoplasty etc.)
* Subjects who had prior silicone injections to their face (Botox and/or Restylane are allowed)
* Subjects considered by the investigator to be smokers
* Subjects with ecchymosis and/or edema on the face on day 0, prior to surgery
* Subjects with known (documented) bleeding or coagulation disorders
* Subjects currently being treated with anti-coagulants
* Subjects treated with Aspirin in the last 7 days or use of other Non-steroidal anti-inflammatory drug (NSAIDs) within the last 7 days prior to surgery
* Subjects with vascular disorders, cardiovascular disease, and/or uncontrolled hypertension
* Subjects with diabetes mellitus
* Subjects with a history of Bell´s palsy
* Subjects with connective tissue disorders
* Subjects with documented history of pathologically or pharmacologically induced immune deficiency
* Subjects receiving systemic corticosteroid treatment for a chronic condition within 2 to 30 days prior to the surgery
* Subjects with a known sensitivity to fibrin sealants
* Subjects with a known psychiatric disorder (e.g., depression, obsessive compulsive disorder, anxiety, eating disorders, etc)
* Subjects who have participated in another clinical study within 30 days prior to this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Z Abrams, MD, Study Director — Baxter Healthcare Corporation
Locations (6):
- United States (6):
  - Beverly Hills, California
  - Los Angeles, California
  - Atlanta, Georgia
  - Evans, Georgia
  - Hewlett, New York
  - Chattanooga, Tennessee

REFERENCES:
- [Derived] Hester TR Jr, Gerut ZE, Shire JR, Nguyen DB, Chen AH, Diamond J, Desmond JC, Silvati-Fidell L, Abrams SZ. Exploratory, randomized, controlled, phase 2 study to evaluate the safety and efficacy of adjuvant fibrin sealant VH S/D 4 S-Apr (ARTISS) in patients undergoing rhytidectomy. Aesthet Surg J. 2013 Mar;33(3):323-33. doi: 10.1177/1090820X13477860. PMID 23515377

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 6 clinical sites in the United States, beginning June 2008 and completing in September 2008
Pre-assignment Details: 56 participants were enrolled and screened. 2 were screen failures. 9 were withdrawn prior to randomization (1 due to untoward medical occurrence, 2 due to study site over enrollment, 2 requested withdrawal, 2 had scheduling conflicts, 1 had surgery delayed, 1 missed deadline for enrollment. Therefore, 45 of the 56 enrolled were randomized.
Groups:
- Facelift Participants: One side of the face is treated with FS VH S/D 4; the other side of the face is treated using standard of care.
Period: Overall Study
Arm/Group | Facelift Participants
Started | 45 (Randomized and treated)
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Facelift Participants
Number analyzed (Participants) | 45
Age Continuous [Mean (Standard Deviation); unit: years] | 55.1 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Visual Comparison of Ecchymosis at Postoperative Day 3
Description: Comparison between the FS VH S/D 4 treated side of the face and the side treated using standard of care (SoC) assessed by 5 separate blinded reviewers using standard digital photographs.
Time Frame: Through Postoperative Day 3
Population: Per Protocol. If there is no majority (i.e., 3 or more in agreement) in the outcomes of the visual comparison of both sides of the face from the 5 blinded reviewers then the assessment will not contribute to the analysis.
Measure: Number; unit: participants
Arm/Group | Participants With Less Ecchymosis Treated With FS VH S/D 4 | Participants With Less Ecchymosis Treated With SoC | Participants With Equal Ecchymosis On Both Sides | Participants With No Ecchymosis on Either Side
Number analyzed (Participants) | 28 | 28 | 28 | 28
participants | 5 | 12 | 11 | 0
Statistical Analysis 1: Comparison: Participants With Less Ecchymosis Treated With FS VH S/D 4 vs Participants With Less Ecchymosis Treated With SoC; Test type: Superiority or Other; p = 0.143, McNemar; Difference in Proportions = 0.250, 95% CI [-0.04 to 0.49] — Difference in Proportions = SoC - FS VH S/D 4

2. Secondary Outcome: Visual Comparison of Ecchymosis at Day 1
Description: as for outcome 1
Time Frame: Through Postoperative Day 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Participants With Less Ecchymosis Treated With FS VH S/D 4 | Participants With Less Ecchymosis Treated With SoC | Participants With Equal Ecchymosis On Both Sides | Participants With No Ecchymosis on Either Side
Number analyzed (Participants) | 29 | 29 | 29 | 29
participants | 2 | 11 | 16 | 0
Statistical Analysis 1: Comparison: Participants With Less Ecchymosis Treated With FS VH S/D 4 vs Participants With Less Ecchymosis Treated With SoC; Test type: Superiority or Other; Difference in proportions = 0.310, 90% CI 2-sided [0.12 to 0.48] — Difference in proportions = SoC - FS VH S/D 4

3. Secondary Outcome: Visual Comparison of Ecchymosis at Day 5
Description: as for outcome 1
Time Frame: Through Postoperative Day 5
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Participants With Less Ecchymosis Treated With FS VH S/D 4 | Participants With Less Ecchymosis Treated With SoC | Participants With Equal Ecchymosis On Both Sides | Participants With No Ecchymosis on Either Side
Number analyzed (Participants) | 27 | 27 | 27 | 27
participants | 5 | 8 | 14 | 0
Statistical Analysis 1: Comparison: Participants With Less Ecchymosis Treated With FS VH S/D 4 vs Participants With Less Ecchymosis Treated With SoC; Test type: Superiority or Other; Difference in proportions = 0.111, 90% CI 2-sided [-0.11 to 0.32] — Difference in proportions = SoC - FS VH S/D 4

4. Secondary Outcome: Visual Comparison of Ecchymosis at Day 7
Description: as for outcome 1
Time Frame: Through Postoperative Day 7
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Participants With Less Ecchymosis Treated With FS VH S/D 4 | Participants With Less Ecchymosis Treated With SoC | Participants With Equal Ecchymosis On Both Sides | Participants With No Ecchymosis on Either Side
Number analyzed (Participants) | 31 | 31 | 31 | 31
participants | 9 | 8 | 14 | 0
Statistical Analysis 1: Comparison: Participants With Less Ecchymosis Treated With FS VH S/D 4 vs Participants With Less Ecchymosis Treated With SoC; Test type: Superiority or Other; Difference in proportions = -0.032, 90% CI 2-sided [-0.24 to 0.18] — Difference in proportions = SoC - FS VH S/D 4

5. Secondary Outcome: Visual Comparison of Ecchymosis at Day 10
Description: as for outcome 1
Time Frame: Through Postoperative Day 10
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Participants With Less Ecchymosis Treated With FS VH S/D 4 | Participants With Less Ecchymosis Treated With SoC | Participants With Equal Ecchymosis On Both Sides | Participants With No Ecchymosis on Either Side
Number analyzed (Participants) | 28 | 28 | 28 | 28
participants | 7 | 7 | 14 | 0
Statistical Analysis 1: Comparison: Participants With Less Ecchymosis Treated With FS VH S/D 4 vs Participants With Less Ecchymosis Treated With SoC; Test type: Superiority or Other; Difference in proportions = 0.000, 90% CI 2-sided [-0.21 to 0.21] — Difference in proportions = SoC - FS VH S/D 4

6. Secondary Outcome: Visual Comparison of Ecchymosis at Day 14
Description: as for outcome 1
Time Frame: Through Postoperative Day 14
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Participants With Less Ecchymosis Treated With FS VH S/D 4 | Participants With Less Ecchymosis Treated With SoC | Participants With Equal Ecchymosis On Both Sides | Participants With No Ecchymosis on Either Side
Number analyzed (Participants) | 26 | 26 | 26 | 26
participants | 5 | 6 | 14 | 1
Statistical Analysis 1: Comparison: Participants With Less Ecchymosis Treated With FS VH S/D 4 vs Participants With Less Ecchymosis Treated With SoC; Test type: Superiority or Other; Difference in proportions = 0.038, 90% CI 2-sided [-0.17 to 0.24] — Difference in proportions = SoC - FS VH S/D 4

7. Secondary Outcome: Difference in Marchac Grades Using A Modified Marchac Scale (MMS) of Ecchymosis Between Two Sides of Face Assessed by 5 Independent, Blinded Reviewers- Day 1
Description: Reviewers used photographs from postoperative Day 1, 3, 5, 7, 10, and 14. Differences are calculated as (SoC Grade) - (FS VH S/D 4 Grade). MMS for Post Rhytidectomy (Facelift) Ecchymosis: Grade 0= No bruising; Grade 1= Barely perceivable (easily hidden with makeup, yellowish color and affects limited area); Grade 2= Present, minimal (yellow color and covers ≤25% of operated area); Grade 3= Moderate (yellow color and covers >25% of operated area, red color, blue color but covers a very small area); Grade 4= Extensive (blue color and covers more than just a very small area, dark purple color)
  The planned and approved Statistical Analysis Plan (SAP) specified a pre-aggregation of the data whereby differences between the two sides of the face were computed first within participants to retain the inherent correlation (pairings) in the measures. Summary statistics and statistical tests were then computed on the differences between the two sides of the face using paired sample tests.
Time Frame: Through Postoperative Day 1
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.0 [-0.2 to 0.0]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.645, Two-sided Wilcoxon paired sample tests; alpha = 10%

8. Secondary Outcome: Difference in Marchac Grades Using A Modified Marchac Scale (MMS) of Ecchymosis Between Two Sides of Face Assessed by 5 Independent, Blinded Reviewers- Day 3
Description: Reviewers used photographs from postoperative Day 1, 3, 5, 7, 10, and 14. Differences are calculated as (SoC Grade) - (FS VH S/D 4 Grade). MMS for Post Rhytidectomy (Facelift) Ecchymosis: Grade 0= No bruising; Grade 1= Barely perceivable (easily hidden with makeup, yellowish color and affects limited area); Grade 2= Present, minimal (yellow color and covers ≤25% of operated area); Grade 3= Moderate (yellow color and covers >25% of operated area, red color, blue color but covers a very small area); Grade 4= Extensive (blue color and covers more than just a very small area, dark purple color)
  The planned and approved SAP specified a pre-aggregation of the data whereby differences between the two sides of the face were computed first within participants to retain the inherent correlation (pairings) in the measures. Summary statistics and statistical tests were then computed on the differences between the two sides of the face using paired sample tests.
Time Frame: Through Postoperative Day 3
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | -0.2 [-0.4 to 0.2]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.103, Two-sided Wilcoxon paired sample tests; alpha = 10%

9. Secondary Outcome: Difference in Marchac Grades Using A Modified Marchac Scale (MMS) of Ecchymosis Between Two Sides of Face Assessed by 5 Independent, Blinded Reviewers- Day 5
Description: as for outcome 8
Time Frame: Through Postoperative Day 5
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.0 [0.0 to 0.2]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.833, Two-sided Wilcoxon paired sample tests; alpha = 10%

10. Secondary Outcome: Difference in Marchac Grades Using A Modified Marchac Scale (MMS) of Ecchymosis Between Two Sides of Face Assessed by 5 Independent, Blinded Reviewers- Day 7
Description: as for outcome 8
Time Frame: Through Postoperative Day 7
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.0 [-0.2 to 0.2]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.501, Two-sided Wilcoxon paired sample tests; alpha = 10%

11. Secondary Outcome: Difference in Marchac Grades Using A Modified Marchac Scale (MMS) of Ecchymosis Between Two Sides of Face Assessed by 5 Independent, Blinded Reviewers- Day 10
Description: as for outcome 8
Time Frame: Through Postoperative Day 10
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.0 [-0.4 to 0.2]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.247, Two-sided Wilcoxon paired sample tests; alpha = 10%

12. Secondary Outcome: Difference in Marchac Grades Using A Modified Marchac Scale (MMS) of Ecchymosis Between Two Sides of Face Assessed by 5 Independent, Blinded Reviewers- Day 14
Description: as for outcome 8
Time Frame: Through Postoperative Day 14
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.0 [-0.2 to 0.4]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.715, Two-sided Wilcoxon paired sample tests; alpha = 10%

13. Secondary Outcome: Difference in Marchac Grades Using A Modified Marchac Scale (MMS) of Ecchymosis Between Two Sides of Face Assessed by a Blinded On-site Evaluator-Day 3
Description: Difference between each side of the face are calculated as (SoC Grade) - (FS VH S/D 4 Grade). MMS for Post Rhytidectomy (Facelift) Ecchymosis: Grade 0= No bruising; Grade 1= Barely perceivable (easily hidden with makeup, yellowish color and affects limited area); Grade 2= Present, minimal (yellow color and covers ≤25% of operated area); Grade 3= Moderate (yellow color and covers >25% of operated area, red color, blue color but covers a very small area); Grade 4= Extensive (blue color and covers more than just a very small area, dark purple color)
  The planned and approved SAP specified a pre-aggregation of the data whereby differences between the two sides of the face were computed first within participants to retain the inherent correlation (pairings) in the measures. Summary statistics and statistical tests were then computed on the differences between the two sides of the face using paired sample tests.
Time Frame: Postoperative Day 3
Population: Per Protocol
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.00 [-3.00 to 1.00]

14. Secondary Outcome: Difference in Marchac Grades of Edema Between Two Sides of Face Assessed by Investigator Day 1
Description: Investigators used the modified Marchac grading to evaluate edema during participant examinations on postoperative Day 1, 3, 5, 7, 10, and 14. The evaluations were performed on both sides of the face. Differences are calculated as Grade for Standard of Care - Grade for FS VH S/D 4.
  Marchac Scale for Post Rhytidectomy (Facelift) Edema: Grade 1= Nil, Grade 2= Minor, Grade 3= Moderate, Grade 4= Marked/unusual amount.
  The planned and approved SAP specified a pre-aggregation of the data whereby differences between the two sides of the face were computed first within participants to retain the inherent correlation (pairings) in the measures. Summary statistics and statistical tests were then computed on the differences between the two sides of the face using paired sample tests.
Time Frame: Through Postoperative Day 1
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 32
Scores on a scale | 0.00 [0.00 to 0.00]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.754, Two-sided Wilcoxon paired sample tests; alpha = 10%

15. Secondary Outcome: Difference in Marchac Grades of Edema Between Two Sides of Face Assessed by Investigator Day 3
Description: Investigators used the modified Marchac grading to evaluate edema during participant examinations on postoperative Day 1, 3, 5, 7, 10, and 14. The evaluations were performed on both sides of the face. Differences are calculated as Grade for Standard of Care - Grade for FS VH S/D 4. Marchac Scale for Post Rhytidectomy (Facelift) Edema: Grade 1= Nil; Grade 2= Minor; Grade 3= Moderate; Grade 4= Marked/unusual amount.
  The planned and approved SAP specified a pre-aggregation of the data whereby differences between the two sides of the face were computed first within participants to retain the inherent correlation (pairings) in the measures. Summary statistics and statistical tests were then computed on the differences between the two sides of the face using paired sample tests.
Time Frame: Through Postoperative Day 3
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.388, Two-sided Wilcoxon paired sample tests; alpha = 10%

16. Secondary Outcome: Difference in Marchac Grades of Edema Between Two Sides of Face Assessed by Investigator Day 5
Description: as for outcome 15
Time Frame: Through Postoperative Day 5
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.234, Two-sided Wilcoxon paired sample tests; alpha = 10%

17. Secondary Outcome: Difference in Marchac Grades of Edema Between Two Sides of Face Assessed by Investigator Day 7
Description: as for outcome 15
Time Frame: Through Postoperative Day 7
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.688, Two-sided Wilcoxon paired sample tests — Two-sided Wilcoxon paired sample tests; alpha = 10%

18. Secondary Outcome: Difference in Marchac Grades of Edema Between Two Sides of Face Assessed by Investigator Day 10
Description: as for outcome 15
Time Frame: Through Postoperative Day 10
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 32
Scores on a scale | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.625, Two-sided Wilcoxon paired sample tests; alpha = 10%

19. Secondary Outcome: Difference in Marchac Grades of Edema Between Two Sides of Face Assessed by Investigator Day 14
Description: as for outcome 15
Time Frame: Through Postoperative Day 14
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.688, Two-sided Wilcoxon paired sample tests; alpha = 10%

20. Secondary Outcome: Difference in Marchac Grades Using A Modified Marchac Scale (MMS) of Ecchymosis Between Two Sides of Face Assessed by Investigator- Day 1
Description: Investigators used MMS during examinations- postoperative Day 1, 3, 5, 7, 10, and 14. Differences are calculated as (SoC Grade) - (FS VH S/D 4 Grade). MMS for Post Rhytidectomy (Facelift) Ecchymosis: Grade 0= No bruising; Grade 1= Barely perceivable (easily hidden with makeup, yellowish color & affects limited area); Grade 2= Present, minimal (yellow color & covers ≤25% of operated area); Grade 3= Moderate (yellow color & covers >25% of operated area, red color, blue color but covers a very small area); Grade 4= Extensive (blue color & covers more than just very small area, dark purple color)
  The planned and approved SAP specified a pre-aggregation of the data whereby differences between the two sides of the face were computed first within participants to retain the inherent correlation (pairings) in the measures. Summary statistics and statistical tests were then computed on the differences between the two sides of the face using paired sample tests.
Time Frame: Through Postoperative Day 1
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 1.000, Two-sided Wilcoxon paired sample tests; alpha = 10%

21. Secondary Outcome: Difference in Marchac Grades Using A Modified Marchac Scale (MMS) of Ecchymosis Between Two Sides of Face Assessed by Investigator- Day 3
Description: as for outcome 20
Time Frame: Through Postoperative Day 3
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.521, Two-sided Wilcoxon paired sample tests; alpha = 10%

22. Secondary Outcome: Difference in Marchac Grades Using A Modified Marchac Scale (MMS) of Ecchymosis Between Two Sides of Face Assessed by Investigator- Day 5
Description: as for outcome 20
Time Frame: Through Postoperative Day 5
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.0 [0.0 to 1.0]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.324, Two-sided Wilcoxon paired sample tests — alpha = 10%

23. Secondary Outcome: Difference in Marchac Grades Using A Modified Marchac Scale (MMS) of Ecchymosis Between Two Sides of Face Assessed by Investigator- Day 7
Description: as for outcome 20
Time Frame: Through Postoperative Day 7
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.661, Two-sided Wilcoxon paired sample tests; alpha = 10%

24. Secondary Outcome: Difference in Marchac Grades Using A Modified Marchac Scale (MMS) of Ecchymosis Between Two Sides of Face Assessed by Investigator- Day 10
Description: as for outcome 20
Time Frame: Through Postoperative Day 10
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 1.000, Two-sided Wilcoxon paired sample tests; alpha = 10%

25. Secondary Outcome: Difference in Marchac Grades Using A Modified Marchac Scale (MMS) of Ecchymosis Between Two Sides of Face Assessed by Investigator- Day 14
Description: as for outcome 20
Time Frame: Through Postoperative Day 14
Population: Per Protocol
Measure: Median (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Facelift Participants; Test type: Superiority or Other; p = 0.699, Two-sided Wilcoxon paired sample tests; alpha = 10%

26. Secondary Outcome: Resolution of Ecchymosis as Assessed by Investigators
Description: Resolution of ecchymosis (grade 0 on the Modified Marchac Scale for ecchymosis (Grade 0 = No bruising at all))
Time Frame: Postoperative Days 1, 3, 5, 7, 10, and 14
Population: Per Protocol
Measure: Number; unit: participants
Arm/Group | Complete Resolution of Ecchymosis With FS VH S/D 4 But Not SoC | Complete Resolution of Ecchymosis With SoC But Not FS VH S/D 4 | Participants With Complete Resolution on Both Sides | Participants With No Resolution on Either Side
Number analyzed (Participants) | 33 | 33 | 33 | 33
participants
  By Day 1 | 0 | 0 | 2 | 31
  By Day 3 | 0 | 0 | 1 | 32
  By Day 5 | 1 | 0 | 0 | 32
  By Day 7 | 1 | 0 | 0 | 32
  By Day 10 | 1 | 0 | 1 | 31
  By Day 14 | 1 | 3 | 7 | 22

27. Secondary Outcome: Resolution of Edema as Assessed by Investigators.
Description: Resolution of edema (grade 1 on the Marchac Scale for Edema (Grade 1 = Nil)
Time Frame: Postoperative Days 1, 3, 5, 7, 10, and 14
Population: Per Protocol
Measure: Number; unit: participants
Arm/Group | Complete Resolution of Edema With FS VH S/D 4 But Not SoC | Complete Resolution of Edema With SoC But Not FS VH S/D 4 | Participants With Complete Resolution on Both Sides | Participants With No Resolution on Either Side
Number analyzed (Participants) | 33 | 33 | 33 | 33
participants
  By Day 1 (n=32) | 3 | 0 | 0 | 29
  By Day 3 (n=33) | 0 | 0 | 0 | 33
  By Day 5 (n=33) | 0 | 0 | 0 | 33
  By Day 7 (n=33) | 1 | 0 | 1 | 33
  By Day 10 (n=32) | 1 | 0 | 1 | 30
  By Day 14 (n=32) | 4 | 2 | 6 | 20

28. Secondary Outcome: Total Volume of Drainage on Each Side of the Face
Time Frame: 24 hours postoperative
Population: Per Protocol
Measure: Median (Full Range); unit: mL
Arm/Group | Standard of Care (SoC) | FS VH S/D 4
Number analyzed (Participants) | 33 | 33
mL | 16 [0.0 to 100.0] | 5 [0.0 to 50.0]
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FS VH S/D 4; Test type: Superiority or Other; p = 0.0010, two-sided paired t-test; alpha = 5%

29. Secondary Outcome: Participants With Hematoma/Seroma
Description: Investigators assessed each side of the face for the presence of hematoma/seroma
Time Frame: Days 0, 1, 3, 5, 7,10, and 14
Population: Per Protocol
Measure: Number; unit: Participants
Arm/Group | Standard of Care (SoC) | FS VH S/D 4
Number analyzed (Participants) | 33 | 33
Participants
  Day 0 | 2 | 0
  Day 1 | 1 | 0
  Day 3 | 2 | 0
  Day 5 | 1 | 0
  Day 7 | 1 | 0
  Day 10 | 2 | 0
  Day 14 | 1 | 0

30. Secondary Outcome: Participants With Hematoma/Seroma During the Study
Description: Investigators assessed each side of the face for the presence of hematoma/seroma
Time Frame: Through Postoperative Day 14 (± 1)
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Participants With Hematoma/Seroma on FS VH S/D 4 Side | Participants With Hematoma/Seroma on SoC Side | Participants With Hematoma/Seroma on Both Sides | Participants With No Hematoma/Seroma on Either Side
Number analyzed (Participants) | 33 | 33 | 33 | 33
participants | 0 | 6 | 0 | 27
Statistical Analysis 1: Comparison: Participants With Hematoma/Seroma on FS VH S/D 4 Side vs Participants With Hematoma/Seroma on SoC Side; Test type: Superiority or Other; p = 0.014, McNemar's test of paired proportions; Alpha = 5%; Difference in proportions = 0.182, 95% CI 2-sided [0.04 to 0.34] — Difference in Proportions = (Number of SoC Participants with Hematoma/Seroma) - (Number of FS VH S/D 4 Participants with Hematoma/Seroma)

31. Secondary Outcome: Differences From Day 0 in Two-Point Discrimination Tests Days 3, 7, 10, 14
Description: Two-point discrimination test performed by investigators to assess nerve regeneration. Testing performed on each side of the face (SoC and FS VH S/D 4). Differences are calculated as: Postoperative Day - Day 0, reported as minimal distance at which participants were able to discern feeling at two distinct points
Time Frame: Postoperative Days 3, 7, 10, and 14
Population: Per protocol
Measure: Median (Full Range); unit: mm
Arm/Group | FS VH S/D 4 - Day3 | SoC - Day 3 | FS VH S/D 4 - Day 7 | SoC - Day 7 | FS VH S/D 4 - Day 10 | SoC - Day 10 | FS VH S/D 4 - Day 14 | SoC - Day 14
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33 | 33 | 33 | 33
mm | 7 [-12 to 48] | 7 [-5 to 44] | 5 [-20 to 48] | 6 [-10 to 59] | 5 [-32 to 37] | 5 [-10 to 45] | 0 [-41 to 38] | 5 [-13 to 39]

32. Secondary Outcome: Differences in Subjects' Assessments of Pain for Each Side of Face (SoC and FS VH S/D 4)
Description: Differences are calculated as (Grade for SoC) - (Grade for FS VH S/D 4). Participants used a 10-point visual analogue scale to complete a pain assessment for each side of their face during each postoperative study visit (Days 1, 3, 5, 7, 10, and 14). The higher the number, the greater the pain experienced, i.e. 10 = worst, 1 = least.
  The planned and approved SAP specified a pre-aggregation of the data whereby differences between the two sides of the face were computed first within participants to retain the inherent correlation (pairings) in the measures. Summary statistics and statistical tests were then computed on the differences between the two sides of the face using paired sample tests.
Time Frame: Days 1, 3, 5, 7,10, and 14
Population: Per Protocol
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale
  Day 1 | 0 [-4 to 3]
  Day 3 | 0 [-4 to 4]
  Day 5 | 0 [-5 to 3]
  Day 7 | 0 [-4 to 2]
  Day 10 | 0 [-1 to 2]
  Day 14 | 0 [-1 to 3]

33. Secondary Outcome: Differences in Subjects' Assessments of Numbness for Each Side of Face (SoC and FS VH S/D 4)
Description: Differences are calculated as (Grade for SoC) - (Grade for FS VH S/D 4). Participants used a 10-point visual analogue scale to complete a numbness assessment for each side of their face during each postoperative study visit (Days 1, 3, 5, 7, 10, and 14). The higher the number, the greater the numbness experienced, i.e. 10 = worst, 1 = least.
  The planned and approved SAP specified a pre-aggregation of the data whereby differences between the two sides of the face were computed first within participants to retain the inherent correlation (pairings) in the measures. Summary statistics and statistical tests were then computed on the differences between the two sides of the face using paired sample tests.
Time Frame: Days 1, 3, 5, 7,10, and 14
Population: Per Protocol
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 33
Scores on a scale
  Day 1 | 0 [-4 to 4]
  Day 3 | 0 [-7 to 4]
  Day 5 | 0 [-2 to 4]
  Day 7 | 0 [-3 to 3]
  Day 10 | 0 [-2 to 2]
  Day 14 | 0 [-3 to 2]

34. Secondary Outcome: Participants' Assessment of Side of Face Preference (SoC and FS VH S/D 4)
Description: Participants compared the levels of bruising on each side of their face and determine if they had a preference for the look of 1 side over another.
Time Frame: Postoperative Days 1, 3, 5, 7, 10, and 14
Population: Per Protocol
Measure: Number; unit: participants
Arm/Group | No Difference | FS VH S/D 4 Looks Better | SoC Looks Better
Number analyzed (Participants) | 33 | 33 | 33
participants
  Day 1 | 5 | 12 | 16
  Day 3 | 1 | 20 | 12
  Day 5 | 2 | 17 | 14
  Day 7 | 2 | 17 | 14
  Day 10 | 5 | 13 | 15
  Day 14 | 5 | 12 | 15

35. Primary Outcome: Incidence of Adverse Events (AEs) Related to Study Product (FS VH S/D 4) Throughout the Study Period
Time Frame: Through Postoperative Day 14 (± 1)
Population: Safety Data Set
Measure: Number; unit: Adverse Events
Arm/Group | Facelift Participants
Number analyzed (Participants) | 45
Adverse Events | 0

ADVERSE EVENTS:
Time Frame: Approximately 16 weeks
Groups:
- Localized to SoC Side of Face: AE was localized to the side of the face which was treated with standard of care.
- Localized to FS VH S/D 4 Side of Face: AE was localized to the side of the face which was treated with FS VH S/D 4.
- Non-localized AEs: AE affected a site other than either side of the face (ie, non-localized AE)
Arm/Group | Localized to SoC Side of Face | Localized to FS VH S/D 4 Side of Face | Non-localized AEs
Serious Adverse Events (participants affected / at risk) | 1/45 | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 10/45 | 3/45 | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Localized to SoC Side of Face (N=45) | Localized to FS VH S/D 4 Side of Face (N=45) | Non-localized AEs (N=45)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Localized to SoC Side of Face (N=45) | Localized to FS VH S/D 4 Side of Face (N=45) | Non-localized AEs (N=45)
Oedema (General disorders) | 3 (4) | 3 (3) | 0 (0)
Haematoma (Vascular disorders) | 7 (7) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs may vary per requirements of the individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 1 year after study completion. Baxter requires a review of results communications (e.g., for confidential information) ≥90 days prior to submission or communication. Baxter may request an additional delay of ≤60 days (e.g., for intellectual property protection)